CLINICAL TRIAL: NCT07402616
Title: Feasibility of 3D ex Vivo Ultrasonography for Post-operative Evaluation of Tumor Margins in Cutaneous Squamous Cell Carcinoma
Brief Title: Ex Vivo Cutaneous SCC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Linnea Langhans, Principal investigator, Rigshospitalet, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Ex vivo cutaneous SCC
Record Dates: First submitted 2026-01-14; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Cutaneous Squamous Cell Carcinoma
Keywords: cSCC; 3D ultrasound; ultrasonography; ex vivo

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 3D Ultrasonography (Experimental)
  Interventions: Diagnostic Test: ex vivo 3D ultrasonography

INTERVENTIONS:
Diagnostic Test: ex vivo 3D ultrasonography — Surgical specimens scanned with 3D ultrasonography

SUMMARY:
This is a prospective study including patients ( ≥ 18 years) referred for surgical treatment of primary cutaneous squamous cell carcinoma at the Department of Plastic Surgery, Rigshospitalet. After written and informed consent, patients will undergo standard surgical excision, followed by ex vivo 3D ultrasonography of the specimen using a 3Sonic device connected to a high-frequency ultrasound machine. This will create 3D ultrasound tomographic scans which will be interpreted by one investigator blinded to histopathology. The investigated outcomes will primarily be the deep margin distance. This will be compared to histopathology, where a pathologist - blinded to the ultrasonography results - will slice the entire specimen parallel to the ultrasound images. A third investigator will then match the histopathology images to the ultrasound images for correlation of the measured deep margins.

ELIGIBILITY:
Inclusion Criteria:

* Adults with primary cutaneous squamous cell carcinoma.

Exclusion Criteria:

* Carcinomas located on the eyelids, vulva, penis, or perianal.
* Tumors with an anticipated excision larger than 60mm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-02-01 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Deep margin distance | Within 10-14 days from enrollment
  The minimum deep margins in each ultrasound or histopathology tumor slide measured in millimeters from the deepest tumor border to the closest deep border of the healthy tissue (if present).

SECONDARY OUTCOMES:
Depth of invasion | Within 10-14 days from enrollment
  Distance perpendicular to the granular layer of the epidermis of the specimen to the deepest point of tumor invasion, measured in millimeters.
Tumor size in 3 dimensions measured in mm with ultrasound and histopathology | Within 10-14 days from enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Todsen, MD, PhD, Study Chair — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided